CLINICAL TRIAL: NCT01572831
Title: A Pilot Study to Evaluate a Procalcitonin-Based Algorithm for Duration of Antibiotic Therapy in Critically Ill Patients
Brief Title: PCT and Clinical Algorithm for Determination of Duration of Antibiotics
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fraser Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FHREB 2011-089
Record Dates: First submitted 2012-04-04; First posted 2012-04-06 (Estimated); Last update posted 2015-05-25 (Estimated); Status verified 2012-04

CONDITIONS: Infection
Keywords: antibiotic cessation rules; procalcitonin; infection; critical care
MeSH Terms: conditions — Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- standard care (No Intervention): Abx will be determined by the managing physician
- experimental arm (Experimental): Abx determined by normalization of PCT and basic clinical parameters
  Interventions: Other: PCT and clinical algorithm for stopping abx

INTERVENTIONS:
Other: PCT and clinical algorithm for stopping abx — In the experimental arm, antibiotics will be stopped based upon the PCT-guided algorithm. This PCT algorithm also incorporates clinical parameters to ensure utmost safety for the patients. These clinical parameters are; resolution of fever (temperature less than 38.3 and greater than 36.0), shock (on no vasopressors), and leukocytosis (<12,000 and >4,000).
  Arms: experimental arm

SUMMARY:
Patients in the ICU whose infection is resolving will be randomized to standard duration of antibiotics compared to duration determined by a combination of a procalcitonin value and a simple evaluation of clinical status.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (19 years and older) treated with ABx for reasons other than prophylaxis within the last 24 hours and who are admitted to a critical care environment.

Exclusion Criteria:

* Declined consent
* Any infection that according to evidence-based guidelines which would usually receive more than 2 weeks of antibiotic therapy including, but not limited to;

  * Infective endocarditis
  * Osteomyelitis
  * Undrained abscess
* Not expected to survive 48 hours
* Immunosuppression (HIV positive, any immunosuppressive medications, any steroid dose, neutrophil count less than 1.0)
* Previously enrolled in this study
* Presently enrolled in a separate study which is felt by study investigators to have biological or clinical process in conflict with this study.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2012-05; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Antibiotic- free days and alive at 14 days after ICU admission | 14 days

SECONDARY OUTCOMES:
mortality at 28 days | 28 days
mortality at 90 days | 90 days
ventilator days at 28 days | 28 days
ICU free days at 28 days | 28 days
relapsed infection | 30 days
rates of CDAD | 30 days
colonization/infection with VRE/MRSA over next 30 days | 30 days
duration of abx in control arm for those with and without formal stewardship programs | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Steven Reynolds, MD, Principal Investigator — University of British Columbia
Locations (1):
- Royal Columbian Hospital, New Westminster, British Columbia, Canada